CLINICAL TRIAL: NCT04004377
Title: Acoustic Neuroma: Assessing the Quality of Life by the Scale PANQOL of Patients Operated or Supervised
Acronym: PANQOL
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2018/39
Record Dates: First submitted 2019-06-28; First posted 2019-07-02 (Actual); Last update posted 2019-07-02 (Actual); Status verified 2019-05

CONDITIONS: Acoustic Neuroma
MeSH Terms: conditions — Neuroma, Acoustic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- acoustic neuroma monitored radiologically: patient with an acoustic neuroma (vestibular schwannoma) with MRI confirmed, unilateral, not yet operated at baseline, aged over 18 years, monitoring by radiology
  Interventions: Other: Scale of quality life
- acoustic neuroma whose treatment is surgical: patient with an acoustic neuroma (vestibular schwannoma or) with MRI confirmed, unilateral, not yet operated at baseline, aged over 18 years, resection surgery planified
  Interventions: Other: Scale of quality life

INTERVENTIONS:
Other: Scale of quality life — The PANQOL scale (Penn Acoustic Neuroma Quality-of-Life) is a specific questionnaire containing 26 items Interviewing 7 areas: hearing, balance, facial expression, anxiety, vitality, pain, and 'general health. The score is encrypted from 0 to 100, and the highest score is a reflection of the best possible quality of life. This score has been translated from French into English and validated according to the reverse translation rules by usual Oddon et al.
  Three questions for this score were added, evaluating quality of life parameters that seem particularly interesting: the first regarding the difficulties in driving, the second questioning the recovery of a "normal" life, and the third assessing difficulties in working life.

SUMMARY:
This study has investigated the quality of life of patients with vestibular schwannoma using this specific scale prospectively, whether treated surgically or monitored.

DETAILED DESCRIPTION:
The PANQOL scale (Penn Acoustic Neuroma Quality-of-Life) is a specific questionnaire containing 26 items Interviewing 7 areas: hearing, balance, facial expression, anxiety, vitality, pain, and 'general health. The score is encrypted from 0 to 100, and the highest score is a reflection of the best possible quality of life. This score has been translated from French into English and validated according to the reverse translation rules by usual Oddon et al.

Three questions for this score were added, evaluating quality of life parameters that seem particularly interesting: the first regarding the difficulties in driving, the second questioning the recovery of a "normal" life, and the third assessing difficulties in working life.

The questionnaires are sent to the patient in the form of a custom web link generated on the online survey platform SurveyMonkey, and integrated into the body of an email sent from the mailbox of the investigator Hospital. There is any identifying or indirectly identifying data on the questionnaire online, guaranteeing protection of the rights of the individual. Only the principal investigator and co-investigator retain the link between the coded identity of persons undergoing research used to associate personal health data and their name (s) and name (s) (correspondence table retained securely to the paper).

ELIGIBILITY:
Inclusion Criteria:

* be in possession of an acoustic neuroma (or vestibular schwannoma) confirmed in MRI, unilateral, unoperated
* Age over 18 years
* patient insured or beneficiary of a social security scheme
* free, informed and express

Exclusion Criteria:

* History of surgery of the angle ponto-cerebellar or otologic
* Neurofibromatosis type 2
* Cons-indication to MRI
* psychiatric pathology
* Pregnant or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited during consultation ear (Multidisciplinary Consultative Meeting) , Neurosurgery of the University Hospital of Bordeaux - be in possession of an acoustic neuroma (or vestibular schwannoma) confirmed in MRI, unilateral, unoperated
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2018-12-05 (Actual); Primary Completion 2020-12-05 (Estimated); Study Completion 2020-12-05 (Estimated)

PRIMARY OUTCOMES:
Score of PANQUOL Questionnaire | Month 1
  The PANQOL scale (Penn Acoustic Neuroma Quality-of-Life) is a specific questionnaire containing 26 items Interviewing 7 areas: hearing, balance, facial expression, anxiety, vitality, pain, and 'general health. The score is encrypted from 0 to 100, and the highest score is a reflection of the best possible quality of life. This score has been translated from French into English and validated according to the reverse translation rules by usual Oddon et al.
Score of PANQUOL Questionnaire | Month 3
  The PANQOL scale (Penn Acoustic Neuroma Quality-of-Life) is a specific questionnaire containing 26 items Interviewing 7 areas: hearing, balance, facial expression, anxiety, vitality, pain, and 'general health. The score is encrypted from 0 to 100, and the highest score is a reflection of the best possible quality of life. This score has been translated from French into English and validated according to the reverse translation rules by usual Oddon et al.
Score of PANQUOL Questionnaire | Month 6
  The PANQOL scale (Penn Acoustic Neuroma Quality-of-Life) is a specific questionnaire containing 26 items Interviewing 7 areas: hearing, balance, facial expression, anxiety, vitality, pain, and 'general health. The score is encrypted from 0 to 100, and the highest score is a reflection of the best possible quality of life. This score has been translated from French into English and validated according to the reverse translation rules by usual Oddon et al.
Score of PANQUOL Questionnaire | Month 12
  The PANQOL scale (Penn Acoustic Neuroma Quality-of-Life) is a specific questionnaire containing 26 items Interviewing 7 areas: hearing, balance, facial expression, anxiety, vitality, pain, and 'general health. The score is encrypted from 0 to 100, and the highest score is a reflection of the best possible quality of life. This score has been translated from French into English and validated according to the reverse translation rules by usual Oddon et al.

CONTACTS AND LOCATIONS:
Overall Officials: Valérie FRANCO-VIDAL, MD, PhD, Principal Investigator — University Hospital, Bordeaux
Locations (1):
- University Hospital, Bordeaux, Bordeaux, France